CLINICAL TRIAL: NCT00875862
Title: Shoulder Adhesive Capsulitis and Ambulatory Continuous Interscalene Nerve Blocks: A Randomized, Triple-Masked, Placebo-Controlled Study
Brief Title: Shoulder Adhesive Capsulitis and Ambulatory Continuous Interscalene Nerve Blocks
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: procedure no longer being done
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Adhesive Capsulitis
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Adhesive Capsulitis; Post-operative Pain
Keywords: UCSD; pain; quality-of-life; range-of-motion; interscalene catheter; nerve block; shoulder; Shoulder Manipulation
MeSH Terms: conditions — Bursitis; Pain, Postoperative; Pain | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. 0.2% Ropivicaine perinueral infusion (Active Comparator): Patients will receive normal standard of care post-manipulation (single-injection brachial plexus nerve block, oral analgesics, and cold therapy). They will then be randomized to 0.2% Ropivicaine attached to the perineural catheter and an infusion will be initiated. The outcome measures will be assessed by study staff on the phone and at regular visits to the surgeon's office.
  Interventions: Procedure: Interscalene catheter with Ropivicaine or normal saline
- 2. Normal Saline perineural infusion (Placebo Comparator): Patients will receive normal standard of care post-manipulation (single-injection brachial plexus nerve block, oral analgesics, and cold therapy). They will then be randomized to normal saline attached to the perineural catheter and an infusion will be initiated. The outcome measures will be assessed by study staff on the phone and at regular visits to the surgeon's office.
  Interventions: Procedure: Interscalene catheter with Ropivicaine or normal saline

INTERVENTIONS:
Procedure: Interscalene catheter with Ropivicaine or normal saline — Patients will be randomized to one of two groups: 0.2% Ropiviciane or normal saline in the infusion pump, following a shoulder manipulation for adhesive capsulitis. The patients will be followed by doctors and study staff to assess pain, range-of-motion and quality-of-life.

SUMMARY:
Research study to determine if putting local anesthetic through a tiny tube next to the nerves that go to the shoulder will improve shoulder range-of-motion following the shoulder procedure performed on the frozen shoulder. It will also help determine if patients have a higher quality-of-life and less pain, require fewer pain pills, experience fewer sleep disturbances, and are more satisfied with their post-procedure pain control.

DETAILED DESCRIPTION:
Primary Specific Aim: To determine if, compared with usual and customary analgesia, the addition of an ambulatory continuous interscalene nerve block will result in increased shoulder abduction following treatment for adhesive capsulitis of the shoulder.

Hypothesis: Following shoulder manipulation under a single-injection interscalene block for adhesive capsulitis, adding a three-day ambulatory continuous interscalene nerve blcok to usual and customary post-manipulation analgesia will result in a significantly greater shoulder abduction improvement the day following the manipulation.

Secondary Specific Aims: To determine if, compared with usual and customary analgesia, the addition of an ambulatory continuous interscalene nerve block will result in an increased quality-of-life and shoulder range-of-motion, as well as a decreased chronic pain following treatment for adhesive capsulitis of the shoulder.

Hypothesis 1: Following shoulder manipulation under a single-injection interscalene blcok for adhesive capsulitis, adding a three-day ambulatory continuous interscalene nerve block to usual and customary post-manipulation analgesia will result in a significantly increased quality-of-life improvement and shoulder range-of-motion compared wiht baseline values after three months.

Hypothesis 2: Following shoulder manipulation undera a single-injection interscalene block for adhesive capsulitis, adding a three-day ambulatory continuous interscalene nerve block to usual and costomary post-manipulation analgesia will result in a significantly decreased chronic pain compared with basedline falues after three months.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing theraputic manipulation for adhesive capsulitis of the shoulder
* age 18 years or older
* accepting a single-injection nerve block for manipulation
* understanding possible perineural infusion-related complications, study protocol, and catheter/pump care
* having caretaker through the first night after manipulation
* having an ASA physical status classification of 1-3

Exclusion Criteria:

* Any contraindications for a CISB
* any physical, mental or medical conditions which, in the opinion of the investigators, may confound quantifying postoperative pain resulting from surgery
* known allergy or other contraindication to the study medications
* pregnancy
* known hepatic or renal insufficiency/disease
* peripheral neuropathy of the surgical extremity
* morbid obesity
* inability to communicate with the investigators and hospital staff
* moderate-to-severe shoulder arthritis
* immunocompromised status of any etiology
* incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Passive glenohumeral abduction, as evaluated using standard goniometry restricting scapular movement in a supine position. The difference in abduction the day following manipulation compared with the pre-manipulation value, expressed as a percentage. | change from baseline: measured immediately prior to manipulation and the morning following the manipulation.

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, M.D., M.S., Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Medical Center, San Diego, California, United States

REFERENCES:
- [Derived] Malhotra N, Madison SJ, Ward SR, Mariano ER, Loland VJ, Ilfeld BM. Continuous interscalene nerve block following adhesive capsulitis manipulation. Reg Anesth Pain Med. 2013 Mar-Apr;38(2):171-2. doi: 10.1097/AAP.0b013e318283475b. No abstract available. PMID 23423135